CLINICAL TRIAL: NCT04640064
Title: Hb A1C Pre and Post Confinement in Latin American Children With Type 1 Diabetes: Dulce Study Group
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General Puyo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0019
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Type1diabetes; Childhood ALL
Keywords: Type 1 diabetes, children, pandemic, HBA1c,
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with type 1 diabetes: Children younger than 17 years with a diagnosis of type 1 diabetes prior to 2018 will be included.

SUMMARY:
A multicenter retrospective observational study among children with type 1 diabetes will be performed. The Objective of this study will be to determine a) the association between the increase in Hba1c in children with type 1 diabetes and confinement due to the COVID 19 pandemic. b) the association between the frequency of patient care during social confinement and the Hba1c values. Different centers from Latin America including Argentina, Peru, Panama, Chile, and Ecuador will participate in this study. Children younger than 17 years with a diagnosis of type 1 diabetes prior to 2018 will be included. Data from the medical records of the participating centers will be collected on the Hb A1c value before and after confinement (6 months completed). The initial (base) value will be taken as a value of HbA1c registered in the patient's Clinical History for the year 2018, 2019, and 2020 pre and post quarantine (Sep-Oct-Nov) 2020, considering compliance with six months of quarantine. Hb A1c should have been performed in the same institution or with the same methods in order to avoid bias.

DETAILED DESCRIPTION:
Research protocol Hb A1C pre and post Confinement in Latin American children with Type 1 Diabetes: Dulce Study Group

The coronavirus disease is caused by an RNA virus called SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) that has spikes on its surface that give a crown appearance under the electron microscope; hence its name.

A recent cluster of pneumonia cases in Wuhan, China, was caused by this new coronavirus, SARS-CoV-2. In December 2019, adults in Wuhan, a central transportation hub in China, began presenting severe pneumonia of unknown origin in local hospitals. On December 31, 2019, China notified the WHO of the outbreak. On January 7, the virus was identified as a SARS-CoV-2. It soon became known that the disease could be transmitted from asymptomatic people and before the onset of symptoms. The infection is acquired either by inhaling drops or touching contaminated surfaces and then touching the nose, mouth, and eyes. The virus is also present in the stool.

The incubation period ranges from 2 to 14 d [median 5 d]. Studies have identified the angiotensin 2 receptor as the receptor through which the virus enters the respiratory mucosa. (1)

What happens in children? Less than 1% of the cases were in children under the age of 10 in Wuhan, China. Unlike adults, most children have a milder clinical course.

One review included 18 studies with 1065 participants with confirmed SARS-CoV-2 infection. All articles were from China, except for one clinical case in Singapore. Most children had mild respiratory symptoms, such as fever, dry cough, fatigue, or asymptomatic. Bronchial thickening and ground-glass opacities were the main radiographic features in symptomatic or asymptomatic patients. There was only 1 case of severe COVID-19 infection, among the articles included, in a 13-month-old baby. None died. In general, pediatric COVID-19 patients had a good prognosis and recovered within 1 to 2 weeks after illness onset. However, children with mild symptoms or asymptomatic can be a source of viral transmission, constituting essential data for the prevention of the pandemic (2,3).

Food insecurity has been linked to the risk of obesity during the pandemic. Individuals are buying ultra-processed, high-calorie foods. As farms dump food like milk and eggs, grocery stores see empty shelves of cookies, chips, sodas and juices, sugary cereals, and ready-to-eat processed foods. Therefore, we anticipate that many individuals will experience high-calorie diets during the pandemic. (4) There is a greater impact in urban areas of an increasingly sedentary lifestyle. The time in front of the screen, video games, etc., is associated with overweight and obesity due to the double problem (longer sedentary time and increased snacks).

What happens in children with diabetes?

Different studies observed a higher risk of morbidity and mortality in older adults who also had diabetes, hypertension, and other risk factors associated with cardiovascular disease. (5)

Diabetes and Pandemic

Latin America includes developing countries with limited resources. In the absence of specific available and approved vaccines and treatments for COVID-19, the only public health tools available are confinement and social distancing (6). These countries implemented strict social restrictions to stop transmission, including complete border closures, restricted movements during day and night, and inter-provincial travel cessation. However, this measure could generate consequences related to the impact of confinement in vulnerable populations such as patients with diabetes mellitus, worsening glycemic control, and increasing the progression of chronic complications related to the disease. Diabetic children had less access to physical activity, healthy eating, and the frequency of face-to-face clinical consultation. Glycosylated hemoglobin (HbA1C) reflects the average blood glucose of the last 3 months. This test is the main tool for assessing glycemic control and is associated with a high predictive value for diabetes complications. It should be performed routinely in all patients with diabetes at the initial evaluation and as part of the follow-up. Measurement every three months determines whether the patients' blood glucose goals have been achieved and maintained (7).

We believe in the need to develop epidemiological tools to measure the impact of the control of diabetes in children by the crisis and improve the understanding of the patterns of diabetes care during the pandemic. We have not found in the references works on the increase of A1c in Latin America before and after confinement. That is why we have developed this protocol.

The Objective of this study will be to determine a) the association between the increase in Hba1c in children with type 1 diabetes and confinement due to the COVID 19 pandemic. b) the association between the frequency of patient care during social confinement and the Hba1c values.

Exclusion Criteria: pregnancy, kidney failure, treatments that alter hydrocarbon metabolism (corticosteroids, chemotherapy, etc.) and chronic iron deficiency pathologies that alter the value of HbA1c.

Material and methods:

A multicenter retrospective observational study among children with type 1 diabetes will be performed. Different centers from Latin America including Argentina, Peru, Panama, Chile, and Ecuador will participate in this study. Children younger than 17 years with a diagnosis of type 1 diabetes prior to 2018 will be included. Data from the medical records of the participating centers will be collected on the Hb A1c value before and after confinement (6 months completed). The initial (base) value will be taken as a value of HbA1c registered in the patient's Clinical History for the year 2018, 2019, and 2020 pre and post quarantine (Sep-Oct-Nov) 2020, considering compliance with six months of quarantine. Hb A1c should have been performed in the same institution or with the same methods in order to avoid bias.

The years will be divided into four-month periods (quartiles). The Hba1c will be recorded in each period. If a patient had two HbA1c values in the same quarter, the values would be averaged. If there is no value of HbA1C in a period, N / A would be placed in the box.

In addition, the impact of confinement on the BMI registered in the semesters (provided that the data is available) 2018, 2019, and 2020 will be completed. The number of consultations made during 2018,2019 and 2020 by each patient will be completed in the corresponding boxes. The number of telemedicine consultations during the quarantine period will be completed.

Children with type 1 diabetes patients from different private and public centers of Latin America will be included. The sampling frame will be their medical records. The sample is made up of clusters (public or private center) in a single stage since all medical records that meet the selection criteria will be reviewed

Other data to be recorded for analysis will be: public or private setting, date of birth, the weight of birth, age, sex, nationality, blood pressure (BP), lipids ( total cholesterol, triglycerides, and HDL-C), vitamin D, date of onset of diabetes, treatment type (traditional, multiple doses, or insulin pump).

For the collection and processing of the data, a spreadsheet will be used and then the data will be uploaded to REDCAP and statistical packages It is important to clarify that the local researcher will prepare the institution's database anonymously and that when the shipment is made, data to other institutions, it will not be possible to individualize patients, to guarantee the anonymity of patients and the confidentiality of their health data. The last four passport numbers will be used.

The χ2 test will be used to compare proportions. When more than 20% of the cells have expected frequencies <5, Fisher will use the exact test. The adjustment to the normal distribution of continuous variables will be evaluated using the Shapiro-Wilks method. When comparing two groups with normal distribution data, the Student's t test will be performed. When the homogeneity of the variances cannot be tested, the Brown Forsyth test will be used. Variables with asymmetric distribution will be log-transformed for analysis.

Several multiple regressions analyses will be performed to examine the relationship between Hb A1c as a dependent variable and BMI, age, sex, frequency of visits, age of diabetes, duration of confinement, lipids, vitamin D, etc. as the independent variables. Values of P <0.05 will be considered significant. The Bonferroni adjustment will be carried out when numerous comparisons are made. Data will be presented as means ± standard deviations. The analyzes will be performed using the statistical software SPSS® (Chicago, IL) version 21.0. A value of p <0.05 will be considered statistically significant

Data collection

DATE NUMBER NAME PASSPORT SEX AGE ( years BIRTH DATE BIRTH WEIGHT (kG) DATE NUMBER OR COSULTATIONS 2018 2019 2020 INSULIN type HBA1C 2018 1 2 3 HBA1C 2019 1 2 3 HBA1C 2020 1 2 3 HEIGHT 2018 1 2 3 WEIGHT 2018 1 2 3 BMI 2018 1 2 3 HEIGHT 2019 1 2 3 WEIGHT 2019 1 2 3 BMI 2019 1 2 3 HEIGHT 2020 1 2 3 WEIGHT 2020 1 2 3 BMI 2020 1 2 3 Cholesterol total mg/dL 2018 2019 2020 HDL-C mg/dL 2018 2019 2020 TRIGLYCERIDES mg/dL 2018 2019 2020 Vitamin D (Nanograms) 2018 2019 2020 SBP 2018 mmHg 1 2 3 SBP 2019 mmHg 1 2 3 SBP 2020 mmHg 1 2 3 DBP 2018 mmHg 1 2 3 DBP 2019 mmHg 1 2 3 DBP 2020 mmHg 1 2 3 Treatment Conventional Treatment Muultiple Doses CSII COVID Positive Yes/NO

References:

1. The Indian Journal of Pediatrics (April 2020) 87(4):281-286 https://doi.org/10.1007/s12098-020-03263-6)
2. N Engl J Med 2020; 382:1663-1665 DOI: 10.1056/NEJMc2005073 & Pediatrics. 2020 Mar 16;e20200702. doi: 10.1542/peds.2020-0702)
3. JAMA Pediatr. Published online April 22, 2020. doi:10.1001/jamapediatrics.2020.146.)
4. Effects of COVID-19 Lockdown on Lifestyle Behaviors in Children with Obesity Living in Verona, Italy: A Longitudinal Study. Obesity (Silver Spring). 2020 Apr 30;10.1002/oby.22861. doi: 10.1002/oby.22861)
5. BMJ 2020;368:m1198 doi: 10.1136/bmj.m1198 (Published 26 March 2020; Bo Li1 • Jing Yang1,2 • Faming Zhao et. Al. Clinical Research in Cardiology (2020) 109:531-538. https://doi.org/10.1007/s00392-020-01626-9).
6. Miller MJ, Loaiza JR, Takyar A, Gilman RH. PLoS Negl Trop Dis. 2020 May; 14(5): e0008265. doi: 10.1371/journal.pntd.0008265.)
7. Ghosal y col, ( S. Ghosal et al. Diabetes & Metabolic Syndrome: Clinical Research & Reviews 14 (2020) 319e323320).

ELIGIBILITY:
Inclusion Criteria: Children with type 1 diabetes younger than 17 years -

Exclusion Criteria: pregnancy, kidney failure, treatments that alter hydrocarbon metabolism (corticosteroids, chemotherapy, etc.), and chronic iron deficiency pathologies that alter the value of HbA1c.

-

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A multicenter retrospective observational study among children with type 1 diabetes will be performed. Different centers from Latin America including Argentina, Peru, Panama, Chile, and Ecuador will participate in this study. Children younger than 17 years with a diagnosis of type 1 diabetes prior to 2018 will be included. Data from the medical records of the participating centers will be collected on the Hb A1c value before and after confinement (6 months completed). The initial (base) value will be taken as a value of HbA1c registered in the patient's Clinical History for the year 2018, 2019, and 2020 pre and post quarantine (Sep-Oct-Nov) 2020, considering compliance with six months of quarantine. Hb A1c should have been performed in the same institution or with the same methods in order to avoid bias.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-22 (Estimated); Primary Completion 2021-03-22 (Estimated); Study Completion 2021-04-22 (Estimated)

PRIMARY OUTCOMES:
Hb A1C pre and post Confinement in Latin American children with Type 1 Diabetes | six months
  The increase in Hba1c in children with type 1 diabetes and confinement due to the COVID 19 pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- Valeria Hirschler, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
We will do our best to be able to share the data with other researchers